CLINICAL TRIAL: NCT02987829
Title: An Open-label Phase 1/2A Study To Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of TRC253, an Androgen Receptor Antagonist, in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: Phase 1/2A Study of TRC253, an Androgen Receptor Antagonist, in Metastatic Castration-resistant Prostate Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 253PC101
Record Dates: First submitted 2016-12-05; First posted 2016-12-09 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Castrate-resistant Prostate Cancer; Adenocarcinoma, Prostate
MeSH Terms: conditions — Adenocarcinoma | interventions — Androgen Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Level 1: TRC253 40 mg daily (Experimental): 40 mg of single-agent TRC253 to be administered as oral capsules once daily
  Interventions: Drug: TRC253
- Dose Level 2: TRC253 80 mg (Experimental): 80 mg of single-agent TRC253 to be administered as oral capsules once daily
  Interventions: Drug: TRC253
- Dose Level 3: TRC253 160 mg (Experimental): 160 mg of single-agent TRC253 to be administered as oral capsules once daily
  Interventions: Drug: TRC253
- Dose Level 4: TRC253 240 mg (Experimental): 240 mg of single-agent TRC253 to be administered as oral capsules once daily
  Interventions: Drug: TRC253
- Dose Level 5: TRC253 280 mg (Experimental): 280 mg of single-agent TRC253 to be administered as oral capsules once daily
  Interventions: Drug: TRC253
- Dose Level 6: TRC253 320 mg (Experimental): 320 mg of single-agent TRC253 to be administered as oral capsules once daily
  Interventions: Drug: TRC253

INTERVENTIONS:
Drug: TRC253 — TRC253 is a high-affinity, small molecule antagonist of the androgen receptor (AR) with inhibitory activity against wild type AR and specific mutated variants of AR. TRC253 blocks AR nuclear translocation as well as AR binding to DNA and is an antagonist of transcription for wild type AR and mutated AR. TRC253 is orally active and does not have agonist activity towards either the wild type or mutated ARs. TRC253 treatment in the Hershberger assay results in complete inhibition of androgen sensitive organ development. TRC253 is efficacious in an LNCaP xenograft model driven by F876L (also known as F877L) mutant AR.
  Other Names: AR Antagonist

SUMMARY:
This is a multi-center, first-in-human, open-label, Phase 1/2A dose-escalation study in which eligible patients with metastatic castration-resistant prostate carcinoma (mCRPC) will receive oral doses of TRC253. The study will be conducted in 2 parts: part 1 (dose escalation) and part 2 (dose expansion).

DETAILED DESCRIPTION:
The patient population consists of men ≥18 years of age with adenocarcinoma of the prostate with metastatic disease. Patients who have not undergone orchiectomy must have serum testosterone levels <50 ng/dL determined within 4 weeks prior to start of study drug, and, if applicable, must have discontinued treatment with first or second generation anti-androgens as specified in the inclusion criteria.

During Part 1 of the study, patients will be assigned sequentially to increasing TRC253 doses. The starting dose of TRC253 is 40 mg once daily, orally. TRC253 doses will be escalated in subsequent cohorts after all patients enrolled in a given cohort have completed the 28-day dose-limiting toxicity (DLT) evaluation period. Dose escalation in Part 1 will follow single-patient dose escalation design until drug-related toxicity occurs. When an initial drug-related toxicity occurs or DLT in a single patient the cohort will be expanded according to 3+3 design rules. Subsequent dose levels will enroll patients based on 3+3 design. At the maximum tolerated dose (MTD) or minimum efficacious dose (MED), up to twelve patients may be enrolled.

Part 2 will consist of two cohorts of initially up to 30 patients (Cohort 1) and up to 30 patients (Cohort 2) to receive TRC253 at the recommended Phase 2 dose (RP2D). The objective of Part 2 is to gather additional information on the safety, pharmacokinetics (PK) and pharmacodynamic (PD) characteristics, and the clinical efficacy of TRC253 in a pre-defined population of patients with metastatic castrate-resistant prostate cancer (mCRPC). Patients enrolled into Part 2 will have received prior treatment with enzalutamide or apalutamide and showed characteristics of acquired resistance based on changes in PSA serum levels. Patients will be centrally screened for the presence of the AR F876L (androgen receptor F876L) mutation from a plasma sample and enrolled into Cohort 1 (AR F876L positive) or Cohort 2 (AR F876L negative). Cohort 2 may be expanded if a specific molecular mechanism sensitizing the mCRPC to TRC253 therapy can be identified retrospectively. Additional patients may be prospectively selected for this specific molecular resistance mechanism and added to Cohort 2 upon recommendation by the medical monitor and Principal Investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Must have received at least 2 prior therapies approved for CRPC; including a prior AR inhibitor (e.g., enzalutamide or apalutamide). (Part 1 only)
2. Must have received enzalutamide or apalutamide. (Note: additional therapies approved for CRPC prior to enzalutamide or apalutamide are allowed.) (Part 2 only)
3. Must have shown clinical characteristics of acquired resistance to enzalutamide or apalutamide defined as: decline in serum PSA ≥50% compared to baseline serum levels by week 12 (±4 weeks) of enzalutamide or apalutamide treatment and before disease progression by PCWG3 PSA criteria, OR disease progression by PCWG3 radiographic criteria. (Part 2 only)

   Parts 1 and 2:
4. Histologically confirmed adenocarcinoma of the prostate with metastatic disease.
5. Male ≥18 years of age.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Prior orchiectomy or serum testosterone levels <50 ng/dL determined within 4 weeks prior to start of study drug.
8. Adequate baseline organ function.
9. Ongoing androgen depletion therapy with a gonadotropin-releasing hormone (GnRH) analog or inhibitor, or orchiectomy (i.e., surgical or medical castration). Note: patients who have not undergone orchiectomy must continue GnRH analog therapy for the duration of this protocol.
10. For patients previously treated with first generation anti-androgens (i.e., flutamide, nilutamide, or bicalutamide), discontinuation of flutamide or nilutamide therapy must occur >4 weeks (>6 weeks for bicalutamide) prior to start of study drug with no evidence of an anti-androgen withdrawal response (i.e., no decline in serum PSA).
11. For patients previously treated with chemotherapy, targeted therapy, immunotherapy, or treatment with an investigational anticancer agent, discontinuation must have occurred ≥2 weeks, or after at least 4 half-lives, whichever is longer, prior to study drug administration. For enzalutamide and apalutamide, the washout period will be at least 3 weeks prior to start of study drug with no evidence of an anti-androgen withdrawal response (i.e., no decline in serum PSA).
12. For patients previously treated with other agents approved for the treatment of prostate cancer (5-α reductase inhibitors, estrogens, others), discontinuation of therapy must have occurred ≥4 weeks prior to start of study drug.
13. Palliative radiotherapy (to bone or soft tissue lesions) must be completed >2 weeks prior to start of study drug.
14. For patients receiving bone-loss prevention treatment (e.g., bisphosphonates or denosumab), the patient must be on stable dose ≥4 weeks prior to start of study drug.
15. A man who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control during the study and for 4 weeks after receiving the last dose of study drug. All men must also not donate sperm during the study and for 90 days after receiving the last dose of study drug.
16. Patient must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
17. Each patient must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study. Consent is to be obtained prior to the initiation of any study-related tests or procedures that are not part of standard-of-care for the patient's disease.

Exclusion Criteria:

1. History of seizures.
2. Previously documented or current brain metastases.
3. Untreated spinal cord compression.
4. Positive test result for human immunodeficiency virus.
5. History of clinically significant cardiovascular disease including.
6. Active or chronic hepatitis B or hepatitis C as demonstrated by hepatitis B surface antigen positivity and/or anti- hepatitis C virus positivity, respectively. Patients with clinically active or chronic liver disease, including liver cirrhosis of Child-Pugh class C, are also excluded.
7. Second primary malignancy that has not been in remission for greater than 3 years. Exceptions that do not require a 3 year remission include: related non-melanoma skin cancer or resected melanoma in situ.
8. Any serious underlying medical or psychiatric condition (e.g., alcohol or drug abuse), dementia or altered mental status or any issue that would impair the ability of the patient to receive or tolerate the planned treatment, to understand informed consent or that in the opinion of the investigator would contraindicate the patient's participation in the study or that would confound the results of the study.
9. Evidence of active viral, bacterial, or systemic fungal infection requiring systemic treatment within 7 days prior to the first dose of study drug. Patients requiring any systemic antiviral, antifungal, or antibacterial therapy for active infection must have completed treatment no less than 7 days prior to the first dose of study drug.
10. Known allergies, hypersensitivity, or intolerance to TRC253 or its excipients.
11. Enrollment in another interventional study.
12. Major surgery (e.g., requiring general anesthesia) within 3 weeks before screening, or has not fully recovered from prior surgery (i.e., unhealed wound), or surgery planned during the time the patient is expected to participate in the study. Note: patients with planned surgical procedures to be conducted under local anesthesia may participate.
13. Plan to father a child while enrolled in this study or within 90 days after the last dose of study drug.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Freddo, MD, Study Director — Tracon Pharmaceuticals Inc.
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Honor Health, Scottsdale, Arizona
  - University of California at Los Angeles, Santa Monica, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579

RESULTS

PARTICIPANT FLOW:
Groups:
- 40 mg TRC253/Daily; 80 mg TRC253/Daily; 160 mg TRC253/Daily; 240 mg TRC253/Daily; 280 mg TRC253/Daily; 320 mg TRC253/Daily: Single-agent TRC253 to be administered as oral capsules once daily.
Period: Overall Study
Arm/Group | 40 mg TRC253/Daily | 80 mg TRC253/Daily | 160 mg TRC253/Daily | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily
Started | 1 | 1 | 2 | 7 | 51 | 10
Completed | 1 | 1 | 2 | 7 | 51 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg TRC253/Daily | 80 mg TRC253/Daily | 160 mg TRC253/Daily | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily | Total
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 51 | 10 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 2 | 12 | 5 | 19
  >=65 years | 1 | 1 | 2 | 5 | 39 | 5 | 53
Age, Continuous [Mean (Full Range); unit: Years] | 80 [80 to 80] | 65 [65 to 65] | 78 [75 to 81] | 68 [56 to 79] | 73 [56 to 90] | 67 [58 to 81] | 72 [56 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 2 | 7 | 51 | 10 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Race/Ethnicity: Black or African American | 0 | 0 | 0 | 0 | 5 | 3 | 8
  Race/Ethnicity: White | 1 | 1 | 1 | 6 | 42 | 6 | 57
  Race/Ethnicity: Other (Patient declined to answer) | 0 | 0 | 1 | 0 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2 | 7 | 51 | 10 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experience Dose Limiting Toxicities by Dose Level
Description: The trial began with single patient dose escalation rules. If 1 of 1 patients at a given dose experienced a DLT, the study transitioned to a 3+3 design. If 1 of 3 patients experienced a DLT, the dose level was expanded to 6 patients. The maximum tolerated dose (MTD) would have been exceeded if ≥ 33% of patients experience DLT at a given dose level. DLT occurred when a patient had 1 or more toxicities outlined in the protocol that was considered at least possibly related to TRC253 during the first 5 weeks of study participation in the trial. In addition, any dose level could be expanded to further explore PK (the target PK concentration associated with activity in preclinical models was 335 ng/mL). The number of DLTs by dose cohort have been presented.
Time Frame: 5 weeks
Population: All patients who received at least a portion of a dose of TRC253 are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg TRC253/Daily | 80 mg TRC253/Daily | 160 mg TRC253/Daily | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 51 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: 280 mg TRC253/Daily; Determination of the maximum tolerated dose; Test type: Other; One dose limiting toxicity occurred at 320 mg daily of grade 3 QTc prolongation therefore the 280 mg dose was determined to be the maximum tolerated dose and selected as the phase 2 dose

2. Secondary Outcome: Number of Participants With a Serum Prostate-specific Antigen (PSA) Response According to Prostate Cancer Working Group (PCWG3) Criteria
Description: Serum prostate-specific antigen (PSA) response according to Prostate Cancer Working Group (PCWG3) criteria is defined as at least a 50% decrease in PSA from baseline confirmed at least 4 weeks later
Time Frame: 12 weeks
Population: Patients with a baseline PSA and at least 1 on study PSA that were confirmed at least 4 weeks later.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg TRC253/Daily | 80 mg TRC253/Daily | 160 mg TRC253/Daily | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 51 | 10
Participants | 0 | 0 | 1 | 0 | 3 | 1

3. Secondary Outcome: Maximum Change in QTcF
Description: Maximum change in QTcF from baseline by dose level
Time Frame: 18 months
Population: Patients who received at least a portion of a dose of TRC253 with a baseline ECG and at least 1 on study ECG.
Measure: Mean (Full Range); unit: msec
Arm/Group | 40 mg TRC253/Daily | 80 mg TRC253/Daily | 160 mg TRC253/Daily | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily
Number analyzed (Participants) | 1 | 0 | 1 | 7 | 50 | 8
msec | 9 [9 to 9] |  | 22 [22 to 22] | 44.62 [32 to 64] | 37.56 [0 to 77] | 42.63 [5 to 93]

4. Secondary Outcome: Percent Change From Baseline in Standard Uptake Value (SUV) to Assess TRC253 Receptor Occupancy
Description: To confirm the recommended phase 2 dose (RP2D), patients at select dose levels will undergo positron emission tomography scan (PET) scans using fluoro-5alpha-dihydrotestosterone (FDHT), a radiopharmaceutical specifically designed to image binding to androgen receptor (AR). Imaging occurred at one center under their existing investigational new drug application (IND) and institutional protocol. A negative change from baseline in the standard uptake value indicate a decrease in metabolic activity of the tumor and indicate increased receptor occupancy of TRC253.
Time Frame: 4 Weeks
Population: TRC253 4 week FDHT-PET response mean SUV based on the 5 hottest lesions (uncorrected)
Measure: Mean (Full Range); unit: Percent Change from Baseline
Arm/Group | 40 mg TRC253/Daily | 80 mg TRC253/Daily | 160 mg TRC253/Daily | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily
Number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 2
Percent Change from Baseline |  |  | -34.1 [-34.1 to -34.1] | -2.81 [-37.32 to 31.71] | 27.78 [27.78 to 27.78] | -45.88 [-57.32 to -34.43]

5. Secondary Outcome: Median Time to Progression by Dose Level
Description: Preliminary anti-tumor effects of TRC253 as assessed by median time to progression by Prostate Cancer Working Group 3 (PCWG3) criteria by dose level
Time Frame: 18 months
Population: In order to be eligible for efficacy analysis patients must have had a baseline CT scan and at least 1 on study CT scan.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- 40 mg TRC253/Daily Dose Levels Combined; 80 mg TRC253/Daily Dose Levels Combined; 160 mg TRC253/Daily Dose Levels Combined; 240 mg TRC253/Daily; 280 mg TRC253/Daily; 320 mg TRC253/Daily: Single-agent TRC253 to be administered as oral capsules once daily.
Arm/Group | 40 mg TRC253/Daily Dose Levels Combined | 80 mg TRC253/Daily Dose Levels Combined | 160 mg TRC253/Daily Dose Levels Combined | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 44 | 8
months | 8.7 [NA to NA] — The upper and lower confidence level cannot be calculated due to the small sample size | 9.5 [NA to NA] — The upper and lower confidence level cannot be calculated due to the small sample size | 4.8 [NA to NA] — The upper and lower confidence level cannot be calculated due to the small sample size | 3.75 [2.01 to NA] — The upper confidence level cannot be calculated due to the small sample size | 4.64 [2.04 to 7.17] | 12.20 [1.91 to NA] — The upper confidence level cannot be calculated due to the small sample size

6. Secondary Outcome: Number of Patients Who Achieved the Target Concentration of TRC253 at Steady State
Description: Determine the number of patients who achieved the target concentration of TRC253 at steady state (target efficacy concentration of 335 ng/mL based on preclinical models).
Time Frame: 28 days
Population: Patients who received at least 75% of planned continuous daily dosing after 28 days of daily dosing enrolled in part 1 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg TRC253/Daily | 80 mg TRC253/Daily | 160 mg TRC253/Daily | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 4 | 6
Participants | 0 | 0 | 0 | 4 | 4 | 5

ADVERSE EVENTS:
Time Frame: 18 months
Description: Duration of participation +28 days
Arm/Group | 40 mg TRC253/Daily | 80 mg TRC253/Daily | 160 mg TRC253/Daily | 240 mg TRC253/Daily | 280 mg TRC253/Daily | 320 mg TRC253/Daily
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/7 | 1/51 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/2 | 2/7 | 13/51 | 3/10
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/2 | 7/7 | 48/51 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg TRC253/Daily (N=1) | 80 mg TRC253/Daily (N=1) | 160 mg TRC253/Daily (N=2) | 240 mg TRC253/Daily (N=7) | 280 mg TRC253/Daily (N=51) | 320 mg TRC253/Daily (N=10)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intramedullary rod insertion (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg TRC253/Daily (N=1) | 80 mg TRC253/Daily (N=1) | 160 mg TRC253/Daily (N=2) | 240 mg TRC253/Daily (N=7) | 280 mg TRC253/Daily (N=51) | 320 mg TRC253/Daily (N=10)
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 4 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 8 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 5 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 3 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 3 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 8 | 4
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1 | 3 | 14 | 5
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 9 | 6
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 4 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 6 | 3
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 5 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 8 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 7 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 6 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 9 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 3 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 10 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 3 | 1
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 3 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 5 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Corneal neovascularisation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 6 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 4 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Subclavian artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1
Neurogenic Bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Pelvic Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 6 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 0
Vesicocutaneous fistula (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT02987829/Prot_SAP_000.pdf